CLINICAL TRIAL: NCT04670848
Title: Validation of a Contactless Sensor for Sleep Apnea Diagnosis Against Polysomnography
Brief Title: Contactless Detection of Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sleepiz AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PSG-Apnea-Essen
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suspected of suffering from sleep apnea (Experimental)
  Interventions: Device: Sleepiz One+ vs. polysomnography
- Healthy volunteers (Experimental)
  Interventions: Device: Sleepiz One+ vs. polysomnography

INTERVENTIONS:
Device: Sleepiz One+ vs. polysomnography — Simultaneous sleep recording with polysomnography and Sleepiz One+ device

SUMMARY:
In this study the inestigators aim to validate the performance of Sleepiz One+ for sleep apnea detection during routine diagnostic sleep studies. Patients who are prescribed polysomnography study will be asked to participate and undergo a simultaneous sleep recording with radar sensor-based device.

ELIGIBILITY:
Inclusion Criteria:

* Age >18years
* Ability and consent to undergo electrophysiological routine assessment
* Patients suspected to suffer from sleep apnea or any other sleep related disorder

Exclusion Criteria:

* Previous enrollment into the current study,
* Enrollment of the investigator, his/her family members and other dependent persons
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, delirium etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Binary classification of subjects based on their sleep apnea severity (AHI ≥= 15) made by Sleepiz One+, compared to PSG data manually scored by sleep technicians | 1 Night

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schöbel, Prof. Dr. med., Principal Investigator — Universitätsmedizin Essen Ruhrlandklinik
Locations (1):
- Universitätsmedizin Essen Ruhrlandklinik, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gross-Isselmann JA, Eggert T, Wildenauer A, Dietz-Terjung S, Grosse Sundrup M, Schoebel C. Validation of the Sleepiz One + as a radar-based sensor for contactless diagnosis of sleep apnea. Sleep Breath. 2024 Aug;28(4):1691-1699. doi: 10.1007/s11325-024-03057-6. Epub 2024 May 14. PMID 38744804